CLINICAL TRIAL: NCT03462485
Title: Pilot Study on the Effects of Participating in a Dementia-friendly Golf Programme on People With Dementia and Their Informal Caregivers
Brief Title: Pilot Study of the Effects of Playing Golf on People With Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bedfordshire (Other)
Responsible Party: Principal Investigator, Prof David Hewson, Professor of Health and Ageing, University of Bedfordshire
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IHREC820
Record Dates: First submitted 2018-03-02; First posted 2018-03-12 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — GOLF protocol

STUDY DESIGN:
Intervention Model Description: The project will be a randomised controlled trial with a partial crossover. Each condition will be followed for eight weeks, with the crossover occurring after eight weeks for the control group. The intervention group will continue for the full sixteen weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Golf intervention (Experimental): The golf intervention will be an eight-week golf programme in which participants will be taught to play golf in two 150-min sessions each week. Each session will begin with 30 minutes of socialising, then 90 minutes playing golf, followed by another 30 minutes socialising. The golf sessions will progress from putting, to chipping, and then a full swing, with sessions taking place on a nine-hole golf course.
  Interventions: Other: Golf
- Control (No Intervention): Control participants will continue their normal activities.

INTERVENTIONS:
Other: Golf — Eight weeks of twice-daily golf training
  Arms: Golf intervention

SUMMARY:
The research question for this study is whether golf is a suitable physical activity for people with dementia (PWD). It follows a qualitative pilot study in Lincoln where PWD enjoyed the activity and caregivers appreciated the service. Golf combines many desirable elements in a physical activity programme that include being outdoors, social, cognitively challenging, no reaction-time component, and being a typical everyday activity. The length of time that golf sessions last could also offer a potential respite from care for caregivers.

Participants will be people with dementia and their caregivers. Eligibility criteria will include having been clinically diagnosed with dementia, being able to stand on one leg for at least six seconds to ensure participants are able to balance sufficiently well to be able to play golf. The study will be undertaken at The London Shire Golf Club, with the golf training provided by the Golf Trust, which is a charitable foundation experienced in providing golf training to people with a range of different disabilities.

The randomised controlled trial study will last 16 weeks, with a partial crossover design. The experimental group with have two eight-week periods of golf while the control group will have eight weeks without golf, then the golf intervention. There will be two 150-min sessions each week, starting with 30 minutes socialising, then 90 minutes playing golf, then 30 minutes socialising. The golf sessions will progress from putting, to chipping, and then a full swing, with sessions taking place on a nine-hole golf course. Participants will be evaluated before and after each eight-week period for physical function, physical activity level, cognitive function, and quality of life. Their caregivers will also provide information related to the PWD in terms of quality of life and psychopathology in dementia, as well as their own quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with dementia (any dementia)
* Receiving post-diagnostic support
* The capacity to give informed consent
* The physical capacity to play golf as determined by a single-leg stance test of balance

Exclusion Criteria:

* Unable to give informed consent
* Without the physical capacity to play golf, as determined by a single-leg stance test of balance

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-09-30 (Estimated); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 5 minutes
  Quality of life will be assessed using the DEMQOL, which is a 28-item scale that was designed for use with all stages of dementia, and is filled in by the interviewer along with with the participant.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | 10 minutes
  Physical function will be assessed using the SPPB, which consists of three tests to measure balance, walking speed, and muscular performance standing up from a chair.
Assessment of Physical Activity in Frail Older People (APAFOP) | 5 minutes
  Physical activity levels will be recorded using the APAFOP, which uses more common activities in older people such as walking, standing, sitting, and lying, which are given intensity ratings and are more typical of the types of activities of older PWD.
Montreal Cognitive Assessment (MoCA) | 10 minutes
  The MoCA is a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
Caregiver assessment of quality of life (DEMQOL-Proxy) | 5 minutes
  An assessment of the caregiver's impression of the quality of life of the PWD they care for.
The C-DEMQOL will be used to assess the quality of life of caregivers of PWD. Quality of life of caregivers (C-DEMQOL) | 5 minutes
  The C-DEMQOL will be used to assess the quality of life of caregivers of PWD.
Neuropsychiatric Inventory (NPI-Q) | 5 minutes
  Caregivers will complete the short form of the NPI-Q to provide an assessment of neuropsychiatric symptoms and associated caregiver distress.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bedfordshire, Luton, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No